CLINICAL TRIAL: NCT05622708
Title: A Multicenter Study of Secukinumab, With a Randomized Double-blind, Placebo-controlled Withdrawal-retreatment Period, to Evaluate Maintenance of Response in Participants With Non-radiographic Axial Spondyloarthritis Who Achieved Remission
Brief Title: A Study of Secukinumab to Evaluate Maintenance of Response in Participants With Non-radiographic Axial Spondyloarthritis Who Achieved Remission
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457I2401; 2022-001153-23 (EudraCT Number); 2023-509320-17-00 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2022-11-09; First posted 2022-11-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non-radiographic Axial Spondyloarthritis
Keywords: nr-AxSpa; non-radiographic axial Spondyloarthritis; Secukinumab; remission; withdrawal; inflammatory back pain; sacroiliitis; AIN457
MeSH Terms: conditions — Non-Radiographic Axial Spondyloarthritis; Sacroiliitis | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: This phase IV, multicenter study uses a double-blind, placebo-controlled, randomized withdrawal design (Treatment Period 2) preceded by an open label lead-in period (Treatment Period 1).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Period 1 (Experimental): Open-label Secukinumab PFS (prefilled syringe) labeled as AIN457 150mg/1mL
  Interventions: Drug: Secukinumab
- Treatment Period 2 (Experimental): Double-blind Secukinumab and Placebo PFS labeled as AIN457 150mg/1mL/Placebo
  Interventions: Drug: Placebo; Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Treatment Period 1: Open-label secukinumab 150 mg PFS s.c. at baseline, Weeks 1, 2, 3 and 4 followed by administration every four weeks up to Week 52.
  Arms: Treatment Period 1
Drug: Placebo — Treatment Period 2: Double-blind placebo PFS s.c. every 4 weeks from Week 56 to Week 116.
  Arms: Treatment Period 2
Drug: Secukinumab — Treatment Period 2: Double-blind secukinumab 150 mg PFS s.c. every 4 weeks from Week 56 to Week 116.
  Escape re-treatment (during Treatment Period 2): Open-label secukinumab 150 mg PFS s.c.
  Arms: Treatment Period 2

SUMMARY:
This study will establish whether prolonged chronic dosing with secukinumab is needed in participants with Non-radiographic axial spondyloarthritis, (nr-axSpA) who have achieved remission. Remission is defined as Ankylosing Spondylitis Disease Activity Score - C-reactive protein (ASDAS-CRP) Inactive Disease (ID) response (ASDAS-CRP < 1.3). Maintenance of remission on continued secukinumab treatment will be evaluated compared to placebo using a randomized withdrawal design. The primary outcome measure for this study is the proportion of participants remaining flare-free at Week 120.

DETAILED DESCRIPTION:
This study will establish whether prolonged chronic dosing with secukinumab is needed in participants with nr-axSpA who have achieved remission. Remission is defined as Ankylosing Spondylitis Disease Activity Score - C-reactive protein (ASDAS-CRP) Inactive Disease (ID) response Inactive Disease (ID) response (ASDAS-CRP < 1.3). The maintenance of remission on continued secukinumab treatment will be evaluated compared to placebo using a randomized withdrawal design. The primary outcome measure for this study is the proportion of participants remaining flare-free at Week 120.

Study treatment will be as follows:

* Open-label Secukinumab PFS (prefilled syringe) will be labeled as AIN457 150mg/1mL
* Double-blind Secukinumab and Placebo PFS will be labeled as AIN457 150mg/1mL/Placebo.

Study duration will be up to 128 weeks from Baseline.

The treatment duration will be up to 120 weeks with last treatment administration at Week 116.

In the Treatment Period 1 participant will attend a site visit approximately 1 month after Baseline and approximately every 12 weeks thereafter. In the Treatment Period 2 participant will attend site visits approximately every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female participants at least 18 years of age
* Clinical diagnosis of axSpA AND according to ASAS axSpA criteria:

  1. Inflammatory back pain for at least 6 months
  2. Onset before 45 years of age
  3. Sacroiliitis on MRI (magnetic resonance imaging) (as assessed by central reader) with ≥ 1 SpA feature OR HLA-B-27 positive with ≥2 SpA features
* Objective signs of inflammation at screening, evident by either MRI with Sacroiliac Joint inflammation (as assessed by central reader) AND / OR hsCRP > ULN (as defined by the central lab)
* Active axSpA as assessed by total BASDAI ≥ 4 cm (0-10 cm) at baseline.
* Spinal pain as measured by BASDAI question #2 ≥ 4 cm (0-10 cm) at baseline.
* Total back pain as measured by VAS (visual analog scale) ≥ 40 mm (0-100 mm) at baseline.
* Participants should have been on at least 2 different NSAIDs (non-steroidal anti-inflammatory drugs) at the highest recommended dose for at least 4 weeks in total prior to baseline with an inadequate response or failure to respond, or less if therapy had to be withdrawn due to intolerance, toxicity or contraindications.

Exclusion Criteria:

* Participants with radiographic evidence for sacroiliitis, grade ≥ 2 bilaterally or grade ≥ 3 unilaterally (radiological criterion according to the modified New York diagnostic criteria for AS) as assessed by central reader.
* Participants taking high potency opioid analgesics (e.g., methadone, hydromorphone, morphine).
* Previous exposure to secukinumab or any other biologic drug directly targeting IL-17 or IL-17 receptor or previous treatment with immunomodulatory biologic agents including those targeting TNFα (tumor necrosis factor α) (unless participants discontinued the treatment with TNFα inhibitor due to a reason other than efficacy [primary or secondary lack of efficacy, inadequate response] and only after appropriate wash-out period prior to baseline was observed).
* History of hypersensitivity to the study drug or its excipients or to drugs of similar chemical classes.
* Active ongoing inflammatory diseases other than nr-axSpA that might confound the evaluation of the benefit of secukinumab therapy, including uveitis.
* Active inflammatory bowel disease.
* History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2028-04-19 (Estimated); Study Completion 2028-06-13 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants remaining flare-free during Treatment Period 2 | Week 120
  The primary efficacy endpoint is the proportion of participants in the randomized withdrawal population remaining flare-free at Week 120. A flare is defined as ASDAS-CRP ≥ 2.1 at 2 consecutive visits, or ASDAS-CRP > 3.5 at any visit during Treatment Period 2, starting at Week 60.
  Parameters used for ASDAS-CRP include:
  * Spinal pain (BASDAI question 2),
  * Patient's global assessment of disease activity,
  * Peripheral pain/swelling (BASDAI question 3),
  * Duration of morning stiffness (BASDAI question 6)
  * C-reactive protein (CRP) in mg/L

SECONDARY OUTCOMES:
Time to flare during Treatment Period 2 | From Week 56 to Week 120
  A flare is defined as ASDAS-CRP ≥ 2.1 at 2 consecutive visits, or ASDAS-CRP > 3.5 at any visit during Treatment Period 2, starting at Week 60.
Number of participants with Adverse Events | From Baseline to Week 128
  Safety and tolerability demonstrated by assessing:
  - Adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- Belgium (4):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Mons
- Brazil (3):
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
- Colombia (3):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Chía, Cundinamarca
  - Novartis Investigative Site, Bucaramanga, Santander Department
- Czechia (2):
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- France (4):
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Rendsburg
- Hungary (6):
  - Novartis Investigative Site, Székesfehérvár, Fejér
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Veszprém
- Israel (3):
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Verona, VR
- Novartis Investigative Site, Kuala Lumpur, Malaysia
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, Chihuahua City
- Netherlands (2):
  - Novartis Investigative Site, Heerlen, Limburg
  - Novartis Investigative Site, Amsterdam, North Holland
- Philippines (2):
  - Novartis Investigative Site, Makati City, National Capital Region
  - Novartis Investigative Site, Manila
- Poland (6):
  - Novartis Investigative Site, Krakow, Lesser Poland Voivodeship
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Sochaczew
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
- Romania (2):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Bucharest
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Adana, Yuregir
  - Novartis Investigative Site, Konya
- Vietnam (2):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com